CLINICAL TRIAL: NCT03489057
Title: Testing the Efficacy of a Couple-Focused, Tailored mHealth Intervention for Symptom Self-Management Among Men With Prostate Cancer and Their Partners
Brief Title: Efficacy of a Couple-Focused mHealth Symptom Self-management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: LCCC 1713; 1R01NR016990-01A1 (NIH)
Record Dates: First submitted 2018-03-13; First posted 2018-04-05 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
Keywords: symptom; family research; self-management; caregiving; social support; mHealth; healthy behavior; self-efficacy; quality of life; care transition
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Health Resources; Family Characteristics

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator and data collectors will be masked to intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PERC Program (Experimental): Prostate Cancer Education and Resources for Couples (PERC) program. Participants assigned to experimental condition will receive access to the PERC website.
  Interventions: Behavioral: Prostate Cancer Education and Resources for Couples (PERC)
- usual care plus NCI website (Active Comparator): Participants in this usual care plus NCI website group will be automatically directed to the NCI prostate cancer website after logging in to the study website homepage.
  Interventions: Behavioral: usual care plus NCI website

INTERVENTIONS:
Behavioral: Prostate Cancer Education and Resources for Couples (PERC) — PERC uses mHealth technologies to dramatically increase couples' accessibility to posttreatment supportive care whenever and wherever they feel comfortable accessing it. PERC aims to improve QOL for both patients and partners by enhancing positive appraisals of illness and boosting self-efficacy, social support from multiple sources, and healthy behaviors for symptom self-management at home.
  Arms: PERC Program
Behavioral: usual care plus NCI website — The usual care plus NCI website provides generic information about prostate cancer treatment options, research, causes, and statistics; coping resources that are not prostate cancer-specific; support from non-providers via a toll free phone and LiveHelp Online Chat about cancer-related questions, clinical trials, and quitting smoking.
  Arms: usual care plus NCI website

SUMMARY:
In this study, the investigators propose to test the efficacy of a couple-focused, web-based tailored prostate cancer symptom management program, Prostate Cancer Education and Resources for Couples (PERC) in a randomized clinical trial. A two-group (PERC versus National Cancer Institute (NCI) website plus treatment as usual) randomized controlled design will be used, and data will be collected at baseline (T1), 4 (T2), 8 (T3), and 12 months (T4) among 300 patients completing initial treatment for localized prostate cancer and their intimate partners (i.e., 600 participants in total).

DETAILED DESCRIPTION:
This randomized clinical trial aims to test the efficacy of a couple-focused, web-based tailored prostate cancer symptom management program, Prostate Cancer Education and Resources for Couples (PERC). The study participants will include 300 patients completing initial treatment for localized prostate cancer and their intimate partners (i.e., 300 dyads and 600 individuals). After informed consent, we will conduct baseline assessment (T1), randomly assign eligible participants to either PERC or the National Cancer Institute (NCI) website, and then collect data at 4 (T2), 8 (T3), and 12 months (T4) post-T1.

ELIGIBILITY:
Inclusion Criteria:

The eligible patients must

1. be 40 to 75 years of age
2. be within 16 weeks (4 months) after completing initial treatment for localized prostate cancer as confirmed by patient and biopsy pathology report) with curative intent, i.e., surgery or radiotherapy +/- hormonal treatment;
3. have no previous cancer history within the past 2 years and not currently in treatment for cancer, or have a concurrent cancer (excluding non-melanomatous skin cancer);
4. experience prostate cancer-specific and/or general symptoms;
5. have a partner who is willing to participate.

The eligible partners must

1. be 18 years or older
2. be identified as the partner by the patient
3. not have been diagnosed with cancer or receiving treatment for cancer within the past 12 months (non-melanomatous skin cancer diagnosis/treatment is acceptable) so that couples can focus their efforts on managing prostate cancer.

Exclusion Criteria:

Patients and their partners will be excluded from the study if they:

* Do not read and speak English (evidenced by their understanding and responses to screening questions and self-reported ability to read English);
* Have cognitive impairment (assessed by the Short Portable Mental Status Questionnaire).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2022-07-06 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lixin (Lee) Song, RN, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Ma C, Adler RH, Neidre DB, Chen RC, Northouse LL, Rini C, Tan X, Song L. Challenges and Approaches to Recruitment for and Retention in a Dyad-Focused eHealth Intervention During COVID-19: Randomized Controlled Trial. J Med Internet Res. 2024 Dec 3;26:e51877. doi: 10.2196/51877. PMID 39625741
- [Derived] Song L, Nielsen ME, Chen RC, Rini C, Keyserling TC, Idiagbonya E, Fuller GP, Northouse L, Palmer MH, Tan X. Testing the efficacy of a couple-focused, tailored eHealth intervention for symptom self-management among men with prostate cancer and their partners: the study protocol. Trials. 2022 Jan 4;23(1):12. doi: 10.1186/s13063-021-05948-5. PMID 34983621
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 280 patients with newly treated localized prostate cancer and their partner caregivers, with a total of 560 individuals into the study
Pre-assignment Details: All participants completed informed consent and the baseline assessment of quality of life, symptoms, and their stress-coping processes.
Groups:
- Participants Receive PERC: Prostate Cancer Education and Resources for Couples (PERC) program. Participants assigned to the experimental condition will receive access to the PERC website.
  Prostate Cancer Education and Resources for Couples (PERC): PERC uses mHealth technologies to dramatically increase couples' accessibility to posttreatment supportive care whenever and wherever they feel comfortable accessing it. PERC aims to improve QOL for both patients and partners by enhancing positive appraisals of illness and boosting self-efficacy, social support from multiple sources, and healthy behaviors for symptom self-management at home.
- Caregivers of Participants Receive PERC: Prostate Cancer Education and Resources for Couples (PERC) program. Participants assigned to the experimental condition will receive access to the PERC website. Caregivers of participants receive PERC.
  Prostate Cancer Education and Resources for Couples (PERC): PERC uses mHealth technologies to dramatically increase couples' accessibility to posttreatment supportive care whenever and wherever they feel comfortable accessing it. PERC aims to improve QOL for both patients and partners by enhancing positive appraisals of illness and boosting self-efficacy, social support from multiple sources, and healthy behaviors for symptom self-management at home.
- Participants Receive Usual Care: Participants in this usual care plus NCI website group will be automatically directed to the NCI prostate cancer website after logging in to the study website homepage.
  Usual Care Plus NCI website: The usual Care Plus NCI website provides generic information about prostate cancer treatment options, research, causes, and statistics; coping resources that are not prostate cancer-specific; support from non-providers via a toll-free phone and LiveHelp Online Chat about cancer-related questions, clinical trials, and quitting smoking.
- Caregivers of Participants Receive Usual Care: Caregivers of participants receive usual care. Participants in this usual care plus NCI website group will be automatically directed to the NCI prostate cancer website after logging in to the study website homepage.
  Usual Care Plus NCI website: The usual Care Plus NCI website provides generic information about prostate cancer treatment options, research, causes, and statistics; coping resources that are not prostate cancer-specific; support from non-providers via a toll-free phone and LiveHelp Online Chat about cancer-related questions, clinical trials, and quitting smoking.
Period: Overall Study
Arm/Group | Participants Receive PERC | Caregivers of Participants Receive PERC | Participants Receive Usual Care | Caregivers of Participants Receive Usual Care
Started | 141 | 141 | 139 | 139
Completed | 106 | 106 | 115 | 115
Not Completed | 35 | 35 | 24 | 24
Not completed — Lost to Follow-up | 16 | 16 | 14 | 14
Not completed — Withdrawal by Subject | 12 | 12 | 8 | 8
Not completed — Protocol Violation | 7 | 7 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PERC Program | Caregivers of Participants Receive PERC | Participants Receive Usual Care | Caregivers of Participants Receive Usual Care | Total
Number analyzed (Participants) | 141 | 141 | 139 | 139 | 560
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.33 (6.87) | 61.38 (7.23) | 63.10 (6.55) | 60.83 (7.50) | 62.41 (7.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 141 | 0 | 138 | 279
  Male | 141 | 0 | 139 | 1 | 281
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 2 | 2 | 14
  Not Hispanic or Latino | 135 | 135 | 135 | 134 | 539
  Unknown or Not Reported | 2 | 0 | 2 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 1 | 4
  Asian | 1 | 3 | 1 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 28 | 25 | 30 | 28 | 111
  White | 107 | 108 | 108 | 104 | 427
  More than one race | 1 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 2 | 4 | 0 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 141 | 141 | 139 | 139 | 560

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life Over Time as Assessed by Functional Assessment of Cancer Treatment (FACT-G) Scores
Description: The Functional Assessment of Cancer Therapy - General (FACT-G) is used to measure change in quality of life of patient and partner from baseline (T1) to T2 (4 months post-T1), T3 (8-months post-T1), and T4 (12-months post-T1). Change from baseline is the post-Baseline values minus the Baseline value. Functional assessment of Cancer Therapy-General is a 27-item survey which assesses physical, social/family, emotional, and functional well-being on a 5-point Likert scale, with 0 indicating "not at all" and 4 indicating "very much" in response to item questions. The total FACT-G score is calculated as the sum of four sub scores including physical, social/family, emotional, and functional well-being. Total scores range between 0-108. Higher scores indicated better well-being. It has also demonstrated sensitivity to change over time.
Time Frame: Baseline, month 4, 8 and 12
Population: The number reported in the results is based on participants.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline -PERC: Baseline Mean FACT-G Score
- PERC 4-months: The mean FACT-G Score of the participant received PERC at 4 months.
- PERC 8-months: The mean FACT-G Score of the participant received PERC at 8 months.
- PERC 12-months: The mean FACT-G Score of the participant received PERC at 12 months.
- Baseline Usual Care: Mean FACT-G Score of participants receive usual care at baseline.
- Usual Care 4 Months: Mean FACT-G Score of participants receiving usual care at 4 months
- Usual Care 8 Months; Usual Care 12 Months.: Mean FACT-G Score of participants receiving usual care at 8 months.
Arm/Group | Baseline -PERC | PERC 4-months | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care 4 Months | Usual Care 8 Months | Usual Care 12 Months.
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 135
score on a scale | 89.48 (12.92) | 90.54 (12.98) | 90.29 (14.49) | 90.42 (12.58) | 88.38 (14.82) | 90.18 (15.40) | 89.07 (15.39) | 88.07 (16.87)
Statistical Analysis 1: Comparison: Baseline -PERC vs PERC 4-months; Test type: Superiority; p = 0.19, Mixed Models Analysis

2. Secondary Outcome: Change in Pain From Baseline to 4-, 8-, and 12-month Post Baseline as Assessed by Patient-Reported Outcome Measurement Information System (PROMIS) Scores
Description: PROMIS Pain Interference - Short Form 6b is used to measure change in Pain Interference among patients and their partners from Baseline (T1) to T2 (4 months post-T1), T3 (8-mon post-T1), and T4 (12-mon post-T1). Required by PROMIS scoring instrument, for all PROMS measurements, total raw scores are translated into T scores for each participant, where the T score rescales the raw score into a standardized T score with a mean of 50 and a standard deviation (SD) of 10. The pain measures the extent to which patients experience problems with pain over the past 7 days using a 5-point Likert scale. Higher scores reflect greater Pain Interference. The score value ranges between 41-78.3.
Time Frame: Baseline, month 4, 8, and 12
Population: The number reported in the results is based on participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline PERC: Baseline Mean PROMIS Pain Score in PERC group
- PERC 4-months: Mean PROMIS Pain Score in PERC group at 4 months
- PERC 8-months: Mean PROMIS Pain Score of PERC group at 8-months
- PERC 12-months: Mean PROMIS Pain Score of PERC group at 12-months
- Baseline Usual Care: Baseline Mean PROMIS Pain Score of Usual Care Group
- Usual Care 4 Months: Mean PROMIS Pain Score of Usual Care Group at 4 months
- Usual Care 8 Months: Mean PROMIS Pain Score of Usual Care Group at 8 months
- Usual Care 12 Months: Mean PROMIS Pain Score of Usual Care Group at 12 months
Arm/Group | Baseline PERC | PERC 4-months | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care 4 Months | Usual Care 8 Months | Usual Care 12 Months
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 135
score on a scale | 48.88 (9.05) | 48.38 (9.07) | 49.25 (9.33) | 48.37 (8.00) | 49.68 (9.55) | 48.53 (9.12) | 50.09 (10.34) | 50.34 (9.77)

3. Secondary Outcome: Change in Fatigue From Baseline to 4-, 8-, and 12-month Post Baseline as Assessed by The Functional Assessment of Cancer Therapy - General (FACT-G) Scores
Description: FACT-G is used to measure the change in the quality of life of patients and partners from baseline (T1) to T2 (4 months post-T1), T3 (8 months post-T1), and T4 (12 months post-T1). Change from baseline is the post-baseline values minus the Baseline value. Functional Assessment of Cancer Therapy-General is a 27-item survey that assesses physical, social/family, emotional, and functional well-being on a 5-point Likert scale, with 0 indicating "not at all" and 4 indicating "very much" in response to item questions. The total FACT-G score is calculated as the sum of four sub-scores including physical, social/family, emotional, and functional well-being. Total scores range between 0-108. Higher scores indicated better well-being. It has also demonstrated sensitivity to change over time.
Time Frame: Baseline, month 4, 8, and 12
Population: The number reported in the results is based on participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline PERC: Baseline Mean PROMIS Fatigue Score PERC group
- PERC 4-months: PERC group Mean PROMIS Fatigue Score at 4-months
- PERC 8-months: Mean PROMIS Fatigue Score of PERC group at 8-months
- PERC 12-months: Mean PROMIS Fatigue Score of PERC group at 12-months
- Baseline Usual Care: Baseline Mean PROMIS Fatigue Score at Usual Care
- Usual Care - 4 Months: Mean PROMIS Fatigue Score of usual care group at 4 months
- Usual Care -8 Moths: Mean PROMIS Fatigue Score of usual care group at 8 months
- Usual Care -12 Months: Mean PROMIS Fatigue Score of usual care group at 12 months
Arm/Group | Baseline PERC | PERC 4-months | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care - 4 Months | Usual Care -8 Moths | Usual Care -12 Months
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 135
score on a scale | 46.99 (9.40) | 45.78 (9.57) | 47.02 (9.94) | 45.77 (9.05) | 48.44 (9.57) | 47.38 (9.79) | 48.57 (9.96) | 48.94 (9.26)

4. Secondary Outcome: Change in Sleep Disturbance From Baseline to 4-, 8-, and 12-month Post Baseline as Assessed by PROMIS Scores
Description: PROMIS Sleep Disturbance Short Form 8b is used to examine change in sleep quality of patients and their partners from Baseline (T1) to T2 (4 months post T1), T3 (8-months post-T1), and T4 (12-months post-T1). Required by the PROMIS scoring instrument, for all PROMS measurements, total raw scores are translated into T scores for each participant, where the T score rescales the raw score into a standardized T score with a mean of 50 and a standard deviation (SD) of 10. The sleep disturbance sub-scale measured the extent to which participants experienced sleep disturbance over the past 7 days using a 5-point Likert scale. Higher scores reflect greater sleep disturbance. Score value ranges between 28.9-76.5.
Time Frame: Baseline, month 4, 8, and 12
Population: The number reported in the results is based on participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline PERC: Baseline Mean PROMIS Sleep Disturbance Score of PERC Group
- PERC 4-months: Mean PROMIS Sleep Disturbance Score of PERC Group at 4-months
- PERC 8-months: Mean PROMIS Sleep Disturbance Score of PERC Group at 8-months
- PERC 12-months: Mean PROMIS Sleep Disturbance Score of PERC Group at 12-months
- Baseline Usual Care: Baseline Mean PROMIS Sleep Disturbance Score of Usual Care Group
- Usual Care 4-months: Mean PROMIS Sleep Disturbance Score of Usual Care Group at 4-months
- Usual Care 8-months: Mean PROMIS Sleep Disturbance Score of Usual Care Group at 8-months
- Usual Care 12-months: Mean PROMIS Sleep Disturbance Score of Usual Care Group at 12-months
Arm/Group | Baseline PERC | PERC 4-months | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care 4-months | Usual Care 8-months | Usual Care 12-months
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 135
units on a scale | 48.82 (9.73) | 48.54 (9.22) | 48.58 (9.26) | 47.43 (9.10) | 49.96 (9.47) | 50.08 (10.26) | 49.59 (9.84) | 49.79 (10.01)

5. Secondary Outcome: Change in Anxiety From Baseline to 4-, 8-, and 12-month Post Baseline as Assessed by PROMIS-Emotional Distress-Anxiety Short Form
Description: PROMIS-Emotional Distress-Anxiety Short Form 7a is used to examine change in anxiety among patients and their partners from Baseline (T1) to T2 (4 months post T1), T3 (8-months post-T1), and T4 (12-months post-T1). For all PROMS measurements, total raw scores are translated into T scores for each participant, where the T score rescales the raw score into a standardized T score with a mean of 50 and a standard deviation (SD) of 10. The anxiety sub-scale of the PROMIS item bank measures the extent to which participants experience anxiety symptoms over the past 7 days using a 5-point Likert scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with the total scores range from 36.3 to 82.7 with higher scores reflect higher anxiety.
Time Frame: Baseline, month 4, 8, and 12
Population: The number reported in the results is based on participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PERC Baseline: Baseline Mean PROMIS-Emotional Distress-Anxiety Score of PERC Group
- PERC 4-months: Mean PROMIS-Emotional Distress-Anxiety Score of PERC Group at 4-months
- PERC 8-months: Mean PROMIS-Emotional Distress-Anxiety Score of PERC Group at 8-months
- PERC 12-months: Mean PROMIS-Emotional Distress-Anxiety Score of PERC Group at 12 months
- Baseline Usual Care: Baseline Mean PROMIS-Emotional Distress-Anxiety Score of Usual Care Group
- Usual Care 4-months: Mean PROMIS-Emotional Distress-Anxiety Score of Usual Care Group at 4-months
- Usual Care 8-months: Mean PROMIS-Emotional Distress-Anxiety Score of Usual Care Group at 8-months
- Usual Care 12-months: Mean PROMIS-Emotional Distress-Anxiety Score of Usual Care Group at 12-months
Arm/Group | PERC Baseline | PERC 4-months | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care 4-months | Usual Care 8-months | Usual Care 12-months
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 135
score on a scale | 45.15 (8.27) | 44.46 (8.12) | 44.32 (8.50) | 44.11 (7.95) | 46.09 (9.40) | 48.04 (9.13) | 48.53 (9.20) | 46.83 (8.95)

6. Secondary Outcome: Change in Depression From Baseline to 4-, 8-, and 12-month Post Baseline as Assessed by PROMIS-Emotional Distress-Depression
Description: PROMIS-Emotional Distress-Depression Short From 8b is used to measure the change in depression scores among patients from Baseline (T1) to T2 (4 months post T1), T3 (8-months post-T1), and T4 (12-months post-T1). Required by the PROMIS scoring instrument, for all PROMIS measurements, total raw scores are translated into T scores for each participant, where the T score rescales the raw score into a standardized T score with a mean of 50 and a standard deviation (SD) of 10. The depression sub-scale of the PROMIS item bank measures the extent to which participants experience depressive symptoms in the past 7 days using a 5-point Likert scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with the total scores range from 24.7 to 63.5 with higher scores indicate greater depressive symptoms.
Time Frame: Baseline, month 4, 8, and 12
Population: The number reported in the results is based on participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline PERC: Baseline Mean PROMIS-Emotional Short Form 8b Score of PERC Group
- PERC 4-months: Mean PROMIS-Emotional Short Form 8b Score of PERC Group at 4-months
- PERC 8-months: Mean PROMIS-Emotional Short Form 8b Score of PERC Group at 8-months
- PERC 12-months: Mean PROMIS-Emotional Short Form 8b Score of PERC Group at 12 -months
- Baseline Usual Care: Mean PROMIS-Emotional Short Form 8b Score of Usual Care Group at baseline
- Usual Care at 4 Months: Mean PROMIS-Emotional Short Form 8b Score of Usual Care Group at 4 months
- Usual Care 8 Months: Mean PROMIS-Emotional Short Form 8b Score of Usual Care Group at 8 months
- Usual Care 12 Months: Mean PROMIS-Emotional Short Form 8b Score of Usual Care Group at 12 month
Arm/Group | Baseline PERC | PERC 4-months | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care at 4 Months | Usual Care 8 Months | Usual Care 12 Months
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 135
score on a scale | 56.50 (7.31) | 56.31 (6.97) | 57.28 (7.16) | 56.54 (7.85) | 56.92 (7.68) | 56.48 (7.89) | 56.66 (7.46) | 56.63 (8.37)

7. Secondary Outcome: Change in Expanded Prostate Cancer Index Composite Short Form (EPIC 26) Urinary Symptom Score (Patient Only)
Description: Urinary symptom scores change by time were measured using patients' self-assessed urinary symptoms subscale of the Expanded Prostate Cancer Index Composite Short Form (EPIC 26) which is designed to evaluate patient urinary function and bother after prostate cancer treatment. EPIC26 was used at Baseline (T1) to T2 (4 months post-T1), T3 (8 months post-T1), and T4 (12 months post-T1). EPIC26 evaluates patients' functional and symptom-specific issues, including urinary, bowel, sexual, and hormonal symptoms and bother. The patient self-report contains 26 items, and the score range is 0-100. Higher scores represent fewer prostate cancer symptoms and better prostate cancer-related quality of life.
Time Frame: Baseline, month 4, 8, and 12
Population: Subjects completed the study assessment at a time point.The number reported participant flow is the dyad with the intention-to-treat principle. Each dyad contains one patient and one partner.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline PERC: PERC Group Baseline Mean PERC/NCI Score
- 4-months PERC Group: PERC Group Mean PERC/NCI Score at 4-months
- PERC 8-months: PERC Group Mean PERC/NCI Score at 8-months
- PERC 12-months: PERC Group Mean PERC/NCI Score at 12-months
- Baseline Usual Care: Usual Care Group Baseline Mean PERC/NCI Score
- Usual Care 4-months: Usual Care Group Mean PERC/NCI Score at 4-months
- Usual Care 8-months: Usual Care Group Mean PERC/NCI Score at 8-months
- Usual Care 12-months: Usual Care Group Mean PERC/NCI Score at 12-months
Arm/Group | Baseline PERC | 4-months PERC Group | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care 4-months | Usual Care 8-months | Usual Care 12-months
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 115
score on a scale | 67.50 (20.45) | 79.25 (16.41) | 82.58 (16.18) | 80.62 (15.99) | 68.14 (19.25) | 79.23 (16.28) | 80.98 (14.74) | 80.75 (17.47)

8. Secondary Outcome: Change in Expanded Prostate Cancer Index Composite Short Form (EPIC 26) Bowel Symptom Score (Patient Only)
Description: Bowel symptom scores change by time and were measured using patients' self-assessed bowel symptoms subscale of the Expanded Prostate Cancer Index Composite Short Form (EPIC 26) which is designed to evaluate patient function and bother after prostate cancer treatment. EPIC was used at Baseline (T1) to T2 (4 months post-T1), T3 (8 months post-T1), and T4 (12 months post-T1). EPIC26 evaluates patients' functional and symptom-specific issues, including urinary, bowel, sexual, and hormonal symptoms and bother. The patient self-report contains 26 items, and the score range is 0-100. Higher scores represent fewer prostate cancer symptoms and better prostate cancer-related quality of life.
Time Frame: Baseline, month 4, 8, and 12
Population: Subjects completed the study assessment at a time point. The number reported participant flow is the dyad with the intention-to-treat principle. Each dyad contains one patient and one partner.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline PERC | 4-months PERC Group | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care 4-months | Usual Care 8-months | Usual Care 12-months
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 115
score on a scale | 91.90 (14.21) | 93.89 (14.76) | 94.20 (10.77) | 95.23 (10.05) | 90.03 (13.86) | 93.23 (12.70) | 93.62 (13.52) | 92.44 (13.03)

9. Secondary Outcome: Change in Expanded Prostate Cancer Index Composite Short Form (EPIC 26) Sexual Symptom Score (Patients Only)
Description: Sexual symptom scores change by time were measured using patients' self-assessed sexual symptoms subscale of the Expanded Prostate Cancer Index Composite Short Form (EPIC 26) which is designed to evaluate patient function and bother after prostate cancer treatment. EPIC was used at Baseline (T1) to T2 (4 months post T1), T3 (8-months post-T1), and T4 (12-months post-T1). EPIC26 evaluates patients' functional and symptom-specific issues, including urinary, bowel, sexual, and hormonal symptoms and bother. The patient self-report contains 26 items, and the score range is 0-100. Higher scores represent fewer prostate cancer symptoms and better prostate cancer-related quality of life.
Time Frame: Baseline, month 4, 8, and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline PERC | 4-months PERC Group | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care 4-months | Usual Care 8-months | Usual Care 12-months
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 115
score on a scale | 22.96 (24.13) | 24.98 (26.73) | 27.65 (26.30) | 28.20 (29.39) | 21.51 (25.64) | 27.40 (27.11) | 27.06 (24.36) | 32.11 (26.32)

10. Secondary Outcome: Change in Expanded Prostate Cancer Index Composite Short Form (EPIC 26) Hormonal Symptom Score (Patient Only)
Description: Hormonal symptom scores change by time were measured using patients' self-assessed hormonal subscale of the Expanded Prostate Cancer Index Composite Short Form (EPIC 26) which is designed to evaluate patient function and bother after prostate cancer treatment. EPIC was used at Baseline (T1) to T2 (4 months post-T1), T3 (8 months post-T1), and T4 (12 months post-T1). EPIC26 evaluates patients' functional and symptom-specific issues, including urinary, bowel, sexual, and hormonal symptoms and bother. The patient self-report contains 26 items, and the score range is 0-100. Higher scores represent fewer prostate cancer symptoms and better prostate cancer-related quality of life.
Time Frame: Baseline, month 4, 8, and 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline PERC | 4-months PERC Group | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care 4-months | Usual Care 8-months | Usual Care 12-months
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 115
score on a scale | 87.57 (14.19) | 85.24 (18.09) | 86.69 (13.86) | 89.41 (11.25) | 85.62 (15.74) | 87.44 (14.47) | 86.95 (15.02) | 86.13 (16.20)

11. Secondary Outcome: Change in Expanded Prostate Cancer Index Composite Short Form (EPIC 26) Urine Symptom Score (Partners Only)
Description: Urinary symptom scores change by time were measured using caregiver assessed urinary symptoms subscale of the 4-item caregiver version of the Expanded Prostate Cancer Index Composite Short Form which is designed to assess how much of a bother/burden patients' prostate cancer symptoms were for the partners themselves. EPIC-caregiver was used Baseline (T1) to T2 (4 months post-T1), T3 (8 months post-T1), and T4 (12 months post-T1). The partner reported how patients' urinary and bowel, sexual, and hormonal symptoms bothered the caregivers. The score range is 0-100. Higher scores represent fewer bother partners reported and better prostate cancer-related quality of life.
Time Frame: Baseline, month 4, 8, and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline PERC: Baseline Mean PERC/NCI Score in PERC Group
- PERC 4-months: Mean PERC/NCI Score at 4-months in PERC Group
- PERC 8-months: Mean PERC/NCI Score at 8-months in PERC Group
- PERC 12-months: Mean PERC/NCI Score at 12-months in PERC Group
- Baseline Usual Care: Baseline Mean PERC/NCI Score in Usual Care Group
- Usual Care 4months: Mean PERC/NCI Score in Usual Care Group at 4 months
- Usual Care - 8 Months: Mean PERC/NCI Score in Usual Care Group at 8 months
- Usual Care -12 Months: Mean PERC/NCI Score in Usual Care Group at 12 months
Arm/Group | Baseline PERC | PERC 4-months | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care 4months | Usual Care - 8 Months | Usual Care -12 Months
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 115
score on a scale | 76.95 (30.19) | 86.03 (21.28) | 90.44 (17.42) | 86.88 (23.19) | 78.60 (26.51) | 87.62 (19.88) | 86.70 (25.99) | 83.05 (26.27)

12. Secondary Outcome: Change in Expanded Prostate Cancer Index Composite Short Form (EPIC 26) Bowel Symptom (Partners Only)
Description: Bowel symptom scores change by time were measured using caregiver-assessed bowel symptoms subscale of the 4-item caregiver version of the Expanded Prostate Cancer Index Composite Short Form which is designed to assess how much of a bother/burden patients' prostate cancer symptoms were for the partners themselves. EPIC-caregiver was used Baseline (T1) to T2 (4 months post T1), T3 (8 months post-T1), and T4 (12 months post-T1). The partner reported how patients' urinary and bowel, sexual, and hormonal symptoms bothered the caregivers. The score range is 0-100. Higher scores represent fewer bother partners reported and better prostate cancer-related quality of life.
Time Frame: Baseline, month 4, 8, and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline PERC | PERC 4-months | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care 4months | Usual Care - 8 Months | Usual Care -12 Months
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 115
score on a scale | 91.13 (20.73) | 96.78 (9.79) | 97.79 (9.47) | 95.00 (13.43) | 92.45 (16.93) | 96.00 (14.09) | 94.15 (17.46) | 92.05 (17.59)

13. Secondary Outcome: Change in Expanded Prostate Cancer Index Composite Short Form (EPIC 26) Hormonal Symptom Score Partners Only)
Description: Hormonal symptom scores change by time were measured using caregiver-assessed hormonal subscale of the 4-item caregiver version of the Expanded Prostate Cancer Index Composite Short Form which is designed to assess how much of a bother/burden patients' prostate cancer symptoms were for the partners themselves. EPIC-caregiver was used Baseline (T1) to T2 (4 months post T1), T3 (8-months post-T1), and T4 (12 months post-T1). The partner reported how patients' urinary and bowel, sexual, and hormonal symptoms bothered the caregivers. The score range is 0-100. Higher scores represent fewer bother partners reported and better prostate cancer-related quality of life.
Time Frame: Baseline, month 4, 8, and 12
Population: Subjects completed the study assessment at a time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline PERC | PERC 4-months | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care 4months | Usual Care - 8 Months | Usual Care -12 Months
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 115
score on a scale | 76.42 (30.29) | 77.23 (31.04) | 73.53 (37.91) | 75.31 (31.45) | 76.98 (28.56) | 73.75 (32.05) | 73.40 (33.95) | 80.40 (27.19)

14. Secondary Outcome: Change in Expanded Prostate Cancer Index Composite Short Form (EPIC 26) Sexual Symptom Score Partners Only)
Description: Sexual symptom scores change by time were measured using caregiver assessed sexual symptoms subscale of the 4-item caregiver version of the Expanded Prostate Cancer Index Composite Short Form which is designed to assess how much of a bother/burden patients' prostate cancer symptoms were for the partners themselves. EPIC-caregiver was used Baseline (T1) to T2 (4 months post T1), T3 (8 months post-T1), and T4 (12 months post-T1). The partner reported how patients' urinary and bowel, sexual, and hormonal symptoms bothered the caregivers. The score range is 0-100. Higher scores represent fewer bother partners reported and better prostate cancer-related quality of life.
Time Frame: Baseline, month 4, 8, and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline PERC | PERC 4-months | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care 4months | Usual Care - 8 Months | Usual Care -12 Months
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 115
score on a scale | 65.11 (38.26) | 66.16 (36.12) | 64.06 (34.74) | 61.56 (36.44) | 63.22 (39.64) | 60.86 (37.82) | 66.67 (38.06) | 65.23 (36.24)

15. Secondary Outcome: Change in Self-efficacy Scores From Baseline to 4-, 8-, and 12-month Post Baseline as Assessed by the Lewis Cancer Self-Efficacy Scale
Description: The Lewis Cancer Self-Efficacy will be used to measure change in patient and partner feelings of self-efficacy in dealing with the patient's cancer diagnosis and treatment from Baseline (T1) to T2 (4 months post T1), T3 (8-months post-T1), and T4 (12-months post-T1). Change from baseline is the post-Baseline values minus the Baseline value. Patients will rate statements about how confident they feel on a scale from 1 to 10, where higher scores indicate higher self-efficacy.
Time Frame: Baseline, month 4, 8, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | PERC Program | Usual Care Plus NCI Website
Number analyzed (Participants) | 282 | 278
score on a scale
  Score change between T2 and T1 | 0.48 (0.75) | -0.75 (0.74)
  Score change between T3 and T1 | -0.90 (0.80) | -0.76 (0.76)
  Score change between T4 and T1 | -1.00 (0.82) | -1.94 (0.79)
Statistical Analysis 1: Comparison: PERC Program vs Usual Care Plus NCI Website; Test type: Superiority; p = 0.48, Mixed Models Analysis

16. Secondary Outcome: Change in Informational Support Scores From Baseline to 4-, 8-, and 12-month Post Baseline as Assessed by PROMIS-Informational Support Short Form
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 8a is a National Institute of Health-funded initiative to develop and validate patient-reported outcomes (PROs) for clinical research and practice. PROMISE is a set of measures that evaluates and monitors physical, mental, and social health. It uses a 5-point Likert scale. The scoring process involved collecting PROMIS data from participants and calculating the PROMIS score as the sum of responses to each question. Then Health Measures Scoring Service was used to calculate the PROMIS T-score - the standardized score. Specifically, PROMIS uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population (T-scores have a mean of 50 and a standard deviation (SD) of 10). On the T-score metric: A score of 40 is one SD lower than the mean of the reference population; A score of 60 is one SD higher than the mean of the reference population.
Time Frame: Baseline, month 4, 8, and 12
Population: Subjects completed the study assessment at a time point. The number reported in the results participant flow is the dyad with the intention-to-treat principle. Each dyad contains one patient and one partner.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PERC Baseline: Baseline Mean PROMIS Informational Support Short Form 8a Score in PERC Group
- PERC 4-months: Mean PROMIS Informational Support Short Form 8a Score of PERC group at 4-months
- PERC 8-months: Mean PROMIS Informational Support Short Form 8a Score at 8-months
- PERC 12-months: Mean PROMIS Informational Support Short Form 8a Score at 12-months
- Baseline Usual Care: Baseline Mean PROMIS Informational Support Short Form 8a Score in Usual Care Group
- Usual Care -4 Months: Mean PROMIS Informational Support Short Form 8a Score of Usual Care group at 4-months
- Usual Care -8 Months: Mean PROMIS Informational Support Short Form 8a Score of Usual Care group at 8-months
- Usual Care -12 Months: Mean PROMIS Informational Support Short Form 8a Score of Usual Care group at 12 -months
Arm/Group | PERC Baseline | PERC 4-months | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care -4 Months | Usual Care -8 Months | Usual Care -12 Months
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 115
score on a scale | 57.24 (8.52) | 57.29 (7.82) | 58.27 (8.44) | 57.52 (8.80) | 57.07 (7.76) | 57.02 (8.87) | 57.21 (8.77) | 57.17 (9.23)

17. Secondary Outcome: Change in Instrumental Support Scores From Baseline to 4-, 8-, and 12-month Post Baseline as Measured by PROMIS Instrumental Support-Short Form 8a
Description: as for outcome 16
Time Frame: Baseline, month 4, 8, and 12
Population: as for outcome 16
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Baseline PERC: Baseline Mean PROMIS Instrumental Support Short Form 8a Score in PERC group
- PERC 4-months: Mean PROMIS Instrumental Support Short Form 8a Score at 4-months in PERC group
- PERC 8-months: Mean PROMIS Instrumental Support Short Form 8a Score at 8-months in PERC group
- PERC 12-months: Mean PROMIS Instrumental Support Short Form 8a Score at 12-months in PERC group
- Baseline Usual Care: Baseline Mean PROMIS Instrumental Support Short Form 8a Score in Usual Care group
- Usual Care -4 Months: Mean PROMIS Instrumental Support Short Form 8a Score at 4-months in Usual Care group
- Usual Care -8 Months: Mean PROMIS Instrumental Support Short Form 8a Score at 8-months in Usual Care group
- Usual Care -12 Months: Mean PROMIS Instrumental Support Short Form 8a Score at 12-months in Usual Care group
Arm/Group | Baseline PERC | PERC 4-months | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care -4 Months | Usual Care -8 Months | Usual Care -12 Months
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 115
score on a scale | 60.38 (6.05) | 60.59 (5.84) | 60.30 (6.45) | 61.22 (6.07) | 60.81 (5.72) | 60.78 (6.14) | 60.89 (6.15) | 59.74 (7.04)

18. Secondary Outcome: Change in Appraisal of Illness Scores From Baseline to 4-, 8-, and 12-month Post Baseline as Measured by Appraisal of Illness Scale
Description: The appraisal of Illness scale is used to measure changes in perception of prostate cancer and related issues among patients and their partners. The Appraisal of Illness scale is a 20-item measure that uses Likert Scales ranging from 1 to 5 (very false to very true). The score range is 1-5. The higher score indicated a better cognitive appraisal of the illness the patient or partner had. The score is calculated by the Prorated mean scale scores. The formula is prorated scale score =[SUM OF ITEM SCORES]x[N OF ITEMS IN SCALE]/[N OF ITEMS ANSWERED]. Measurements were performed at baseline (T1) to T2 (4 months post T1), T3 (8-months post-T1), and T4 (12-months post-T1). Change from baseline is the post-baseline values minus the baseline value. Higher scores indicate better support.
Time Frame: Baseline, month 4, 8, and 12
Population: Subjects completed the study assessment at a time point.The number reported in the results participant flow is the dyad with the intention-to-treat principle. Each dyad contains one patient and one partner.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline PERC: Baseline Mean The Appraisal of Illness scale Score in PERC group
- PERC 4-months: Mean The Appraisal of Illness scale Score at 4-months n PERC group
- PERC 8-months: Mean The Appraisal of Illness scale Score at 8-months n PERC group
- PERC 12-months: Mean The Appraisal of Illness scale Score at 12-months n PERC group
- Baseline Usual Care: Baseline Mean The Appraisal of Illness scale Score in Usual Care group
- Usual Care 4 Months: Mean The Appraisal of Illness scale Score at 4-months in Usual Care group
- Usual Care 8 Months: Mean The Appraisal of Illness scale Score at 8-months in Usual Care group
- Usual Care 12 Months: Mean The Appraisal of Illness scale Score at 12-months in Usual Care group
Arm/Group | Baseline PERC | PERC 4-months | PERC 8-months | PERC 12-months | Baseline Usual Care | Usual Care 4 Months | Usual Care 8 Months | Usual Care 12 Months
Number analyzed (Participants) | 141 | 113 | 104 | 106 | 139 | 112 | 113 | 115
score on a scale | 3.73 (0.61) | 3.86 (0.73) | 3.83 (0.72) | 3.95 (0.66) | 3.81 (0.70) | 3.86 (0.70) | 3.91 (0.70) | 3.83 (0.72)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: Only Adverse Events that occurred in patient participants were reported. Patient participants' caregivers were not included in adverse event reporting.
Groups:
- PERC Program- Patients Participants: Prostate Cancer Education and Resources for Couples (PERC) program. Participants assigned to experimental condition will receive access to the PERC website.
  Prostate Cancer Education and Resources for Couples (PERC): PERC uses mHealth technologies to dramatically increase couples' accessibility to posttreatment supportive care whenever and wherever they feel comfortable accessing it. PERC aims to improve QOL for both patients and partners by enhancing positive appraisals of illness and boosting self-efficacy, social support from multiple sources, and healthy behaviors for symptom self-management at home.
- Usual Care Plus NCI Website- Patients Participants: Participants in this usual care plus NCI website group will be automatically directed to the NCI prostate cancer website after logging in to the study website homepage.
  Usual care plus NCI website: The usual Care plus NCI website provides generic information about prostate cancer treatment options, research, causes, and statistics; coping resources that are not prostate cancer-specific; support from non-providers via a toll-free phone and LiveHelp Online Chat about cancer-related questions, clinical trials, and quitting smoking.
Arm/Group | PERC Program- Patients Participants | Usual Care Plus NCI Website- Patients Participants
All-Cause Mortality (participants affected / at risk) | 1/141 | 0/139
Serious Adverse Events (participants affected / at risk) | 3/141 | 1/139
Other Adverse Events (participants affected / at risk) | 0/141 | 0/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PERC Program- Patients Participants (N=141) | Usual Care Plus NCI Website- Patients Participants (N=139)
188244007 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 — The patient's cancer had spread.
sudden death (General disorders) | 1 | 0 — The patient had died suddenly while working out at the gym.

LIMITATIONS AND CAVEATS:
1) North Carolina experienced extreme weather events, including storms and flooding (2018, 2019, and 2022), Hurricanes Florence (Category 4, 2018) and Isaias (Category 1, 2020), and Tropical Storm Michael (2018); 2) the control group was exposed to an improved standard of care as the NCI website became substantially more interactive, user-friendly, and sophisticated; 3) the COVID-19 brought ubiquitous online communication and mental distress. All might have affected the study outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT03489057/Prot_SAP_000.pdf